CLINICAL TRIAL: NCT04912245
Title: A Telehealth Advance Care Planning Intervention in Those With Mild Cognitive Impairment or Unrecognized Dementia (Tele Voice)
Brief Title: A Telehealth Advance Care Planning Intervention in Those With Mild Cognitive Impairment or Unrecognized Dementia
Acronym: ACP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00074429; U54AG063546 (NIH)
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2022-07

CONDITIONS: Advance Care Planning; Telemedicine; Mild Cognitive Impairment; Unrecognized Dementia; Dementia
Keywords: Dementia; telehealth; Advance Care Planning; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: This is a pragmatic pilot study where 300 patients with either mild cognitive impairment (MCI) or unrecognized dementia and their care partner (if available) will be approached to participate in a telehealth Advance Care Planning (ACP) visit with a member of their primary care team in hopes of enrolling 94 patients. Patients are still eligible to participate in the study even if a care partner/loved one does not attend the ACP visit with them or if the patient does not have a care partner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth visit (Other): Patients with either MCI or unrecognized dementia and their care partners (if available) will be approached to participate in a telehealth Advance Care Planning (ACP) visit with a member of the patient's primary care team via either telephone or video. Patients without willing or available care partners are still eligible to participate in the study.
  Interventions: Behavioral: Telehealth visit

INTERVENTIONS:
Behavioral: Telehealth visit — Patients with either MCI or unrecognized dementia and their care partners (if available) will be approached to participate in a telehealth Advance Care Planning (ACP) visit with a member of the patient's primary care team via either telephone or video. Patients without willing or available care partners are still eligible to participate in the study.

SUMMARY:
The purpose of this study is to pilot test a telehealth Advance Care Planning (ACP) intervention among those with either mild cognitive impairment (MCI) or unrecognized dementia. Our goal is to pilot-test and evaluate a pragmatic Telehealth ACP intervention among patients with either the diagnosis of mild cognitive impairment (MCI) or unrecognized dementia.

DETAILED DESCRIPTION:
Telehealth has the potential to overcome barriers related to timing and travel restraints and to provide patients and their caregivers with an opportunity to discuss their goals, values, and priorities for their healthcare within their home setting. Recent studies have demonstrated patients' willingness to use telehealth and have shown that it can play an integral role in dementia care management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recognized or probable Mild cognitive impairment (MCI) or mild dementia determined by either ICD10 diagnostic codes or electronic health record (EHR) Risk of Alzheimer's and Dementia Assessment Rule (eRADAR)
* Have decisional capacity according to their primary care physician (PCP) to complete ACP
* Completed visit with their PCP within the past 12 months
* Affiliated with an Accountable Care Organization.
* English-speaking

Exclusion Criteria:

* Moderate to severe hearing loss that would preclude participating in a video or telephone intervention
* No phone number available for patient.
* Lives in a long-term care facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Gabbard, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (7):
- United States (7):
  - Geriatric Medicine-Plaza 1 Davie, Bermuda Run, North Carolina
  - Wake Forest Health Network Family Medicine Conover, Conover, North Carolina
  - WFHN Family Medicine-Premier, High Point, North Carolina
  - Wake Forest Health Network Internal Medicine, Jamestown, North Carolina
  - WFBIK Geriatric Medicine-Kernersville, Kernersville, North Carolina
  - WFHN Family Medicine-Thomasville, Thomasville, North Carolina
  - Geriatric Medicine- Sticht Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayton D, Gardam M, Ward S, Brodaty H, Pritchard E, Earnest A, Krysinska K, Banaszak-Holl J, McNeil J, Ahern S. How Can Quality of Dementia Care Be Measured? The Development of Clinical Quality Indicators for an Australian Pilot Dementia Registry. J Alzheimers Dis. 2020;75(3):923-936. doi: 10.3233/JAD-191044. PMID 32390616
- [Background] Harrison KL, Hunt LJ, Ritchie CS, Yaffe K. Dying With Dementia: Underrecognized and Stigmatized. J Am Geriatr Soc. 2019 Aug;67(8):1548-1551. doi: 10.1111/jgs.15895. Epub 2019 Mar 25. No abstract available. PMID 30908605
- [Background] Mantovani E, Zucchella C, Schena F, Romanelli MG, Venturelli M, Tamburin S. Towards a Redefinition of Cognitive Frailty. J Alzheimers Dis. 2020;76(3):831-843. doi: 10.3233/JAD-200137. PMID 32568197
- [Background] Sugimoto T, Ono R, Kimura A, Saji N, Niida S, Sakai T, Rakugi H, Toba K, Sakurai T. Impact of Cognitive Frailty on Activities of Daily Living, Cognitive Function, and Conversion to Dementia Among Memory Clinic Patients with Mild Cognitive Impairment. J Alzheimers Dis. 2020;76(3):895-903. doi: 10.3233/JAD-191135. PMID 32568192
- [Background] Borda M, G, Soennesyn H, Steves C, J, Osland Vik-Mo A, Pérez-Zepeda M, U, Aarsland D: Frailty in Older Adults with Mild Dementia: Dementia with Lewy Bodies and Alzheimer's Disease. Dement Geriatr Cogn Disord Extra 2019;9:176-183. doi: 10.1159/000496537
- [Background] Gabbard J, Johnson D, Russell G, Spencer S, Williamson JD, McLouth LE, Ferris KG, Sink K, Brenes G, Yang M. Prognostic Awareness, Disease and Palliative Understanding Among Caregivers of Patients With Dementia. Am J Hosp Palliat Care. 2020 Sep;37(9):683-691. doi: 10.1177/1049909119895497. Epub 2019 Dec 19. PMID 31854201
- [Background] Bond WF, Kim M, Franciskovich CM, Weinberg JE, Svendsen JD, Fehr LS, Funk A, Sawicki R, Asche CV. Advance Care Planning in an Accountable Care Organization Is Associated with Increased Advanced Directive Documentation and Decreased Costs. J Palliat Med. 2018 Apr;21(4):489-502. doi: 10.1089/jpm.2017.0566. Epub 2017 Dec 5. PMID 29206564
- [Background] Bischoff KE, Sudore R, Miao Y, Boscardin WJ, Smith AK. Advance care planning and the quality of end-of-life care in older adults. J Am Geriatr Soc. 2013 Feb;61(2):209-14. doi: 10.1111/jgs.12105. Epub 2013 Jan 25. PMID 23350921
- [Background] Mehta A, Kelley AS. Advance Care Planning Codes-Getting Paid for Quality Care. JAMA Intern Med. 2019 Jun 1;179(6):830-831. doi: 10.1001/jamainternmed.2018.8105. No abstract available. PMID 30855636
- [Background] Brinkman-Stoppelenburg A, Rietjens JA, van der Heide A. The effects of advance care planning on end-of-life care: a systematic review. Palliat Med. 2014 Sep;28(8):1000-25. doi: 10.1177/0269216314526272. Epub 2014 Mar 20. PMID 24651708
- [Background] Houben CHM, Spruit MA, Groenen MTJ, Wouters EFM, Janssen DJA. Efficacy of advance care planning: a systematic review and meta-analysis. J Am Med Dir Assoc. 2014 Jul;15(7):477-489. doi: 10.1016/j.jamda.2014.01.008. Epub 2014 Mar 2. PMID 24598477
- [Background] Sinuff T, Dodek P, You JJ, Barwich D, Tayler C, Downar J, Hartwick M, Frank C, Stelfox HT, Heyland DK. Improving End-of-Life Communication and Decision Making: The Development of a Conceptual Framework and Quality Indicators. J Pain Symptom Manage. 2015 Jun;49(6):1070-80. doi: 10.1016/j.jpainsymman.2014.12.007. Epub 2015 Jan 24. PMID 25623923
- [Background] Hammes BJ, Rooney BL, Gundrum JD. A comparative, retrospective, observational study of the prevalence, availability, and specificity of advance care plans in a county that implemented an advance care planning microsystem. J Am Geriatr Soc. 2010 Jul;58(7):1249-55. doi: 10.1111/j.1532-5415.2010.02956.x. PMID 20649688
- [Background] Sellars M, Chung O, Nolte L, Tong A, Pond D, Fetherstonhaugh D, McInerney F, Sinclair C, Detering KM. Perspectives of people with dementia and carers on advance care planning and end-of-life care: A systematic review and thematic synthesis of qualitative studies. Palliat Med. 2019 Mar;33(3):274-290. doi: 10.1177/0269216318809571. Epub 2018 Nov 8. PMID 30404576
- [Background] Sudore RL, Heyland DK, Lum HD, Rietjens JAC, Korfage IJ, Ritchie CS, Hanson LC, Meier DE, Pantilat SZ, Lorenz K, Howard M, Green MJ, Simon JE, Feuz MA, You JJ. Outcomes That Define Successful Advance Care Planning: A Delphi Panel Consensus. J Pain Symptom Manage. 2018 Feb;55(2):245-255.e8. doi: 10.1016/j.jpainsymman.2017.08.025. Epub 2017 Sep 1. PMID 28865870
- [Background] Volhard T, Jessen F, Kleineidam L, Wolfsgruber S, Lanzerath D, Wagner M, Maier W. Advance directives for future dementia can be modified by a brief video presentation on dementia care: An experimental study. PLoS One. 2018 May 24;13(5):e0197229. doi: 10.1371/journal.pone.0197229. eCollection 2018. PMID 29795605
- [Background] Harrison Dening K, Sampson EL, De Vries K. Advance care planning in dementia: recommendations for healthcare professionals. Palliat Care. 2019 Feb 27;12:1178224219826579. doi: 10.1177/1178224219826579. eCollection 2019. PMID 30833812
- [Background] Mitchell SL, Kiely DK, Lipsitz LA. The risk factors and impact on survival of feeding tube placement in nursing home residents with severe cognitive impairment. Arch Intern Med. 1997 Feb 10;157(3):327-32. PMID 9040301
- [Background] Teno JM, Mitchell SL, Kuo SK, Gozalo PL, Rhodes RL, Lima JC, Mor V. Decision-making and outcomes of feeding tube insertion: a five-state study. J Am Geriatr Soc. 2011 May;59(5):881-6. doi: 10.1111/j.1532-5415.2011.03385.x. Epub 2011 May 3. PMID 21539524
- [Background] Mitchell SL, Teno JM, Intrator O, Feng Z, Mor V. Decisions to forgo hospitalization in advanced dementia: a nationwide study. J Am Geriatr Soc. 2007 Mar;55(3):432-8. doi: 10.1111/j.1532-5415.2007.01086.x. PMID 17341248
- [Background] Teno JM, Gruneir A, Schwartz Z, Nanda A, Wetle T. Association between advance directives and quality of end-of-life care: a national study. J Am Geriatr Soc. 2007 Feb;55(2):189-94. doi: 10.1111/j.1532-5415.2007.01045.x. PMID 17302654
- [Background] Givens JL, Prigerson HG, Jones RN, Mitchell SL. Mental health and exposure to patient distress among families of nursing home residents with advanced dementia. J Pain Symptom Manage. 2011 Aug;42(2):183-91. doi: 10.1016/j.jpainsymman.2010.10.259. Epub 2011 Mar 12. PMID 21402461
- [Background] Kiely DK, Givens JL, Shaffer ML, Teno JM, Mitchell SL. Hospice use and outcomes in nursing home residents with advanced dementia. J Am Geriatr Soc. 2010 Dec;58(12):2284-91. doi: 10.1111/j.1532-5415.2010.03185.x. PMID 21143437
- [Background] De Vleminck A, Morrison RS, Meier DE, Aldridge MD. Hospice Care for Patients With Dementia in the United States: A Longitudinal Cohort Study. J Am Med Dir Assoc. 2018 Jul;19(7):633-638. doi: 10.1016/j.jamda.2017.10.003. Epub 2017 Nov 16. PMID 29153752
- [Background] Piers R, Albers G, Gilissen J, De Lepeleire J, Steyaert J, Van Mechelen W, Steeman E, Dillen L, Vanden Berghe P, Van den Block L. Advance care planning in dementia: recommendations for healthcare professionals. BMC Palliat Care. 2018 Jun 21;17(1):88. doi: 10.1186/s12904-018-0332-2. PMID 29933758
- [Background] Bally KW, Krones T, Jox RJ. Advance Care Planning for People with Dementia: The Role of General Practitioners. Gerontology. 2020;66(1):40-46. doi: 10.1159/000500809. Epub 2019 Jun 18. PMID 31212289
- [Background] Farrell TW, Ferrante LE, Brown T, Francis L, Widera E, Rhodes R, Rosen T, Hwang U, Witt LJ, Thothala N, Liu SW, Vitale CA, Braun UK, Stephens C, Saliba D. AGS Position Statement: Resource Allocation Strategies and Age-Related Considerations in the COVID-19 Era and Beyond. J Am Geriatr Soc. 2020 Jun;68(6):1136-1142. doi: 10.1111/jgs.16537. PMID 32374440
- [Background] Block BL, Smith AK, Sudore RL. During COVID-19, Outpatient Advance Care Planning Is Imperative: We Need All Hands on Deck. J Am Geriatr Soc. 2020 Jul;68(7):1395-1397. doi: 10.1111/jgs.16532. Epub 2020 May 14. No abstract available. PMID 32359075
- [Background] Shigekawa E, Fix M, Corbett G, Roby DH, Coffman J. The Current State Of Telehealth Evidence: A Rapid Review. Health Aff (Millwood). 2018 Dec;37(12):1975-1982. doi: 10.1377/hlthaff.2018.05132. PMID 30633674
- [Background] Tousi B. Dementia Care in the Time of COVID-19 Pandemic. J Alzheimers Dis. 2020;76(2):475-479. doi: 10.3233/JAD-200461. PMID 32651326
- [Background] Bossen AL, Kim H, Williams KN, Steinhoff AE, Strieker M. Emerging roles for telemedicine and smart technologies in dementia care. Smart Homecare Technol Telehealth. 2015;3:49-57. doi: 10.2147/SHTT.S59500. Epub 2015 Mar 22. PMID 26636049
- [Background] Guisado-Fernandez E, Blake C, Mackey L, Silva PA, Power D, O'Shea D, Caulfield B. A Smart Health Platform for Measuring Health and Well-Being Improvement in People With Dementia and Their Informal Caregivers: Usability Study. JMIR Aging. 2020 Jul 23;3(2):e15600. doi: 10.2196/15600. PMID 32706650
- [Background] Williams K, Blyler D, Vidoni ED, Shaw C, Wurth J, Seabold D, Perkhounkova Y, Van Sciver A. A randomized trial using telehealth technology to link caregivers with dementia care experts for in-home caregiving support: FamTechCare protocol. Res Nurs Health. 2018 Jun;41(3):219-227. doi: 10.1002/nur.21869. Epub 2018 Mar 5. PMID 29504666
- [Background] Lee E. Do Technology-Based Support Groups Reduce Care Burden Among Dementia Caregivers? A Review. J Evid Inf Soc Work. 2015;12(5):474-87. doi: 10.1080/15433714.2014.930362. Epub 2015 Mar 20. PMID 25794367
- [Background] Malmgren Fange A, Schmidt SM, Nilsson MH, Carlsson G, Liwander A, Dahlgren Bergstrom C, Olivetti P, Johansson P, Chiatti C; TECH@HOME Research Group. The TECH@HOME study, a technological intervention to reduce caregiver burden for informal caregivers of people with dementia: study protocol for a randomized controlled trial. Trials. 2017 Feb 9;18(1):63. doi: 10.1186/s13063-017-1796-8. PMID 28183323
- [Background] Hatcher-Martin JM, Adams JL, Anderson ER, Bove R, Burrus TM, Chehrenama M, Dolan O'Brien M, Eliashiv DS, Erten-Lyons D, Giesser BS, Moo LR, Narayanaswami P, Rossi MA, Soni M, Tariq N, Tsao JW, Vargas BB, Vota SA, Wessels SR, Planalp H, Govindarajan R. Telemedicine in neurology: Telemedicine Work Group of the American Academy of Neurology update. Neurology. 2020 Jan 7;94(1):30-38. doi: 10.1212/WNL.0000000000008708. Epub 2019 Dec 4. PMID 31801829
- [Background] Gabbard J, Pajewski NM, Callahan KE, Dharod A, Foley KL, Ferris K, Moses A, Willard J, Williamson JD. Effectiveness of a Nurse-Led Multidisciplinary Intervention vs Usual Care on Advance Care Planning for Vulnerable Older Adults in an Accountable Care Organization: A Randomized Clinical Trial. JAMA Intern Med. 2021 Mar 1;181(3):361-369. doi: 10.1001/jamainternmed.2020.5950. PMID 33427851
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Barnes DE, Zhou J, Walker RL, Larson EB, Lee SJ, Boscardin WJ, Marcum ZA, Dublin S. Development and Validation of eRADAR: A Tool Using EHR Data to Detect Unrecognized Dementia. J Am Geriatr Soc. 2020 Jan;68(1):103-111. doi: 10.1111/jgs.16182. Epub 2019 Oct 14. PMID 31612463
- [Background] Wilkinson T, Ly A, Schnier C, Rannikmae K, Bush K, Brayne C, Quinn TJ, Sudlow CLM; UK Biobank Neurodegenerative Outcomes Group and Dementias Platform UK. Identifying dementia cases with routinely collected health data: A systematic review. Alzheimers Dement. 2018 Aug;14(8):1038-1051. doi: 10.1016/j.jalz.2018.02.016. Epub 2018 Apr 3. PMID 29621480
- [Background] Nakagawa S, Johnson PCD, Schielzeth H. The coefficient of determination R2 and intra-class correlation coefficient from generalized linear mixed-effects models revisited and expanded. J R Soc Interface. 2017 Sep;14(134):20170213. doi: 10.1098/rsif.2017.0213. Epub 2017 Sep 13. PMID 28904005
- [Background] Allore HG, Goldfeld KS, Gutman R, Li F, Monin JK, Taljaard M, Travison TG. Statistical Considerations for Embedded Pragmatic Clinical Trials in People Living with Dementia. J Am Geriatr Soc. 2020 Jul;68 Suppl 2(Suppl 2):S68-S73. doi: 10.1111/jgs.16616. PMID 32589276
- [Background] Dong H, Robison LL, Leisenring WM, Martin LJ, Armstrong GT, Yasui Y. Estimating the burden of recurrent events in the presence of competing risks: the method of mean cumulative count. Am J Epidemiol. 2015 Apr 1;181(7):532-40. doi: 10.1093/aje/kwu289. Epub 2015 Feb 17. PMID 25693770
- [Background] Rondeau V, Marzroui Y, Gonzalez JR. frailtypack: An R Package for the Analysis of Correlated Survival Data with Frailty Models Using Penalized Likelihood Estimation or Parametrical Estimation. 2012. 2012;47(4):28.
- [Background] Oliveira IR, Molenberghs G, Demetrio CG, Dias CT, Giolo SR, Andrade MC. Quantifying intraclass correlations for count and time-to-event data. Biom J. 2016 Jul;58(4):852-67. doi: 10.1002/bimj.201500093. Epub 2016 Feb 22. PMID 26899931
- See also: Telehealth Survey — https://www.sykes.com/reports/2020-telehealth-survey/
- See also: 2019 Tech Trends and the 50+ — https://doi.org/10.26419/res.00269.001
- See also: Centers for Medicare & Medicaid (2020) Medicare Telemedicine Health Care Provider Fact Sheet — https://www.cms.gov/newsroom/fact-sheets/medicare-telemedicine-health-care-provider-fact-sheet

RESULTS

PARTICIPANT FLOW:
Groups:
- Telehealth Visit-Patients: Patients with either Mild Cognitive Impairment (MCI) or unrecognized dementia and their care partners (if available) will be approached to participate in a telehealth Advance Care Planning (ACP) visit with a member of the patient's primary care team via either telephone or video. Patients without willing or available care partners are still eligible to participate in the study.
  Telehealth visit: Patients with either MCI or unrecognized dementia and their care partners (if available) will be approached to participate in a telehealth Advance Care Planning (ACP) visit with a member of the patient's primary care team via either telephone or video. Patients without willing or available care partners are still eligible to participate in the study.
- Caregivers: Caregivers to Patients
Period: Overall Study
Arm/Group | Telehealth Visit-Patients | Caregivers
Started | 107 | 45
Completed (Caregivers Completed) | 81 | 30
Not Completed | 26 | 15
Not completed — Withdrawal by Subject | 21 | 4
Not completed — Lost to Follow-up | 5 | 11

BASELINE CHARACTERISTICS:
Arm/Group | Telehealth Visit
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 25 Withdrew 16 Lost to Follow
  years
    Patients: number analyzed (Participants) | 107
    Patients | 83.7 (6.5)
    Caregivers: number analyzed (Participants) | 45
    Caregivers | 70.5 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 16 Lost to Follow 25 Withdrew
  Participants
    Patients: number analyzed (Participants) | 107
    Patients: Female | 73
    Patients: Male | 34
    caregivers: number analyzed (Participants) | 45
    caregivers: Female | 36
    caregivers: Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 25 Withdrew 16 Lost to Follow
  Participants
    Patients: number analyzed (Participants) | 107
    Patients: Hispanic or Latino | 4
    Patients: Not Hispanic or Latino | 103
    Patients: Unknown or Not Reported | 0
    Caregivers: number analyzed (Participants) | 45
    Caregivers: Hispanic or Latino | 3
    Caregivers: Not Hispanic or Latino | 42
    Caregivers: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 25 Withdrew 16 Lost to follow
  Participants
    Patients: number analyzed (Participants) | 107
    Patients: American Indian or Alaska Native | 0
    Patients: Asian | 0
    Patients: Native Hawaiian or Other Pacific Islander | 0
    Patients: Black or African American | 18
    Patients: White | 89
    Patients: More than one race | 0
    Patients: Unknown or Not Reported | 0
    Caregivers: number analyzed (Participants) | 45
    Caregivers: American Indian or Alaska Native | 0
    Caregivers: Asian | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0
    Caregivers: Black or African American | 7
    Caregivers: White | 37
    Caregivers: More than one race | 0
    Caregivers: Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patient/Care Partner Agreeing to Participate
Description: Study will measure the amount of patient or patient-care partner dyads who agree to participate.
Time Frame: Baseline to Month 9
Population: 213 Screened - 168 Patients and 45 Caregivers - 152 enrolled (107 Patients and 45 Caregivers)
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Visit
Number analyzed (Participants) | 213
Participants | 152

2. Primary Outcome: Number of Participants With Telehealth Advance Care Planning (ACP) Completed
Description: Study will measure the amount of patients or patient-care partner dyads who complete the ACP telehealth intervention.
Time Frame: month 9
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Visit
Number analyzed (Participants) | 152
Participants | 111

3. Secondary Outcome: Number of Participants With One or More Advance Care Planning (ACP) Discussions
Description: Study will measure the number of ACP discussions documented in the electronic health record.
Time Frame: month 9
Population: 107 enrolled - 26 Withdrawals and Lost To Follows = 81 Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Visit
Number analyzed (Participants) | 81
Participants | 81

4. Secondary Outcome: Number of Participants Who Used One or More Advance Care Planning (ACP) Billing Codes
Description: Study will measure the usage of ACP billing codes (99497 and 99498).
Time Frame: month 9
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Visit
Number analyzed (Participants) | 81
Participants | 78

5. Secondary Outcome: Quality of Advance Care Planning (ACP) Discussion Scores
Description: Discussion quality will be operationalized using a scoring system derived from the ACP Wise documentation program. Score range of 0 (indicating no advance care planning questions answered) to 9 (indicating nine advance care planning questions answered). High-quality ACP discussions will be defined as addressing ≥4 out of 9 core components in the ACP discussion, with 1 point assigned if the following factors were addressed as part of the ACP discussion: Disease understanding, health-related goals, what matters most in their life, important milestones, health-related worries, named surrogate decision-maker, unacceptable states at the end-of-life (e.g. being in a coma, etc.), goals if their health was to worsen, and documentation of code status.
Time Frame: month 9
Population: 107 enrolled - 26 Withdraws and Lost to Follows = 81 Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telehealth Visit
Number analyzed (Participants) | 81
score on a scale | 7.7 (1.7)

ADVERSE EVENTS:
Time Frame: month 9
Groups:
- Telehealth Visit: Patients with either MCI or unrecognized dementia and their care partners (if available) will be approached to participate in a telehealth Advance Care Planning (ACP) visit with a member of the patient's primary care team via either telephone or video. Patients without willing or available care partners are still eligible to participate in the study.
  Telehealth visit: Patients with either MCI or unrecognized dementia and their care partners (if available) will be approached to participate in a telehealth Advance Care Planning (ACP) visit with a member of the patient's primary care team via either telephone or video. Patients without willing or available care partners are still eligible to participate in the study.
  Both Arms/Groups were combined since these were dyad visits - there we zero Adverse Events in the Care Partners Group and one AE in the Participant Group
Arm/Group | Telehealth Visit
All-Cause Mortality (participants affected / at risk) | 1/152
Serious Adverse Events (participants affected / at risk) | 1/152
Other Adverse Events (participants affected / at risk) | 0/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telehealth Visit (N=152)
death (Social circumstances) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT04912245/Prot_SAP_000.pdf